CLINICAL TRIAL: NCT02756767
Title: Assessing the Impact of Electronic Capture of Patient Reported Outcomes in Radiation Oncology
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 24915
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Patients With Lung, Breast, Head and Neck, or Pelvic Malignancies
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Completed subjects: Subjects will complete patient-reported outcomes assessments during and after radiation therapy.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
The goals of this study are to assess the feasibility of weekly administration of site specific patient reported assessments using an electronic platform and to explore the correlation between patient reported outcomes as well as known dosimetric prognostic factors in patients with lung, breast, head and neck, or pelvic malignancies

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer, lung cancer, head and neck cancer, or gynecologic cancer receiving definitive external beam radiotherapy.
* Must be ≥ 18 years of age
* Able to read, write, and speak English in order to complete patient reported outcomes.

Patients will be approached about the study at the time of consultation or at the time of simulation by their treating physicians or by a research coordinator. All patients must sign a study-specific informed consent to participate. All patients, including those who do not choose to consent to the study, will be provided with a short survey to assess health literacy using the eHealth Literacy Scale (eHEALS).

For those not consenting to the study, the survey will be de-identified and will also ask for basic demographic information including age grouping, race, education level, and type of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer, lung cancer, head and neck cancer, or gynecologic cancer receiving definitive external beam radiotherapy.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-04; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Number of Surveys completed | five years

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States